CLINICAL TRIAL: NCT04909255
Title: The Therapeutic Effect of Beta-3 Agonist and Anti-muscarinic Agent on Overactive Bladder Among Sjogren's Syndrome Patient
Brief Title: Beta-3 Agonist and Anti-muscarinic Agent for Sjogren's Syndrome With Overactive Bladder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH109-REC2-200
Record Dates: First submitted 2021-04-21; First posted 2021-06-01 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Sjogren's Syndrome; Overactive Bladder Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — mirabegron; oxybutynin; Tolterodine Tartrate; Solifenacin Succinate; tartaric acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antimuscarinic (Active Comparator): oxybutynin, tolterodine, solifenacin
  Interventions: Drug: oxybutynin, tolterodine, solifenacin
- B3-agonist (Experimental): mirabegron
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — use beta-3 agonist for sjogren syndrome patient
  Other Names: Betmiga
  Arms: B3-agonist
Drug: oxybutynin, tolterodine, solifenacin — use anti-muscarinic agent for patient with overactive bladder syndrome
  Other Names: Ditropan, tartrate, vesicare
  Arms: Antimuscarinic

SUMMARY:
Overactive bladder is more prevalent among the Sjogren syndrome's population compare to the general population. Both anti-muscarinic agent and beta-3 agonist are recommended as second line treatment for overactive bladder syndrome. However, theoretically, undesirable effect of the anti-muscarinic agent such as dry mouth and constipation would make it less suitable for Sjogren syndrome patient with overactive bladder. Therefore, this study is a randomised control study with the aim to evaluate the therapeutic effect of beta-3 agonist and anti-muscarinic agent on overactive bladder among sjogren's syndrome patient.

DETAILED DESCRIPTION:
Overactive bladder(OAB) is a syndrome characterized by the presence of frequency, urgency, nocturia, and with or without urgency urinary incontinence. The reported prevalence of overactive bladder was similar between man and woman. An overactive bladder has been shown to impair the quality of life of the patient. Muscarinic receptors, particularly M2 and M3 receptors were involved in detrusor contraction. Anti-muscarinic receptor drugs, such as oxybutynin and tolterodine are drugs that are currently recommended by both European association of Urology(EAU) and American Urology Association(AUA) guidelines as a second-line treatment for OAB. Beta-3 agonist such as mirabegron is another medication that is commonly used for OAB. Beta-3 agonists increased the bladder capacity of OAB patients without impairing the detrusor contractility.

Sjogren syndrome(Ss) is an autoimmune disease that frequently affects the lacrimal gland and salivary gland causing the patient to have dry mouth and dry eyes. Extraglandular manifestation was also present. Genitourinary manifestation such as frequency, urgency, and vaginal dryness have been reported but not extensively studied. Currently, there is no consensus for the management of these extraglandular manifestations.

Several studies have reported an increasing prevalence of lower urinary tract symptoms in Ss. Detrusor overactivity was the most commonly found based on a small study. A nationwide population-based study in Taiwan has shown that the risk of developing OAB in the Ss population is significantly higher than the control group.

Cholinesterase inhibitors like pilocarpine and muscarinic agonists such as cevimeline are common drugs used to treat dry eyes and dry mouth of Sjogren syndrome while anti-muscarinic drugs are extensively used to treat OAB. Pilocarpine works by increasing acetylcholine concentration in the synaptic junction while cevimeline works as a muscarinic receptor. Whether the increased prevalence of OAB in Ss population is due to the medication itself or due to the disease is not clear. Currently, there is no study investigating the optimal management of lower urinary tract symptoms(LUTS) in Sjogren Syndrome populations.

Objective The objective of this study is to investigate the effect of muscarinic agonists used for Ss on LUTS and the efficacy of beta3 agonists for management OAB in Ss.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sjogren's syndrome AND
* Clinical diagnosis of OAB

Exclusion Criteria:

* Congenital or acquired anatomic abnormalities of the genitourinary tract,
* Uncontrolled severe hypertension >180 mmHg
* Cannot cooperate for voiding diary documentation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Overactive bladder symptom score | 3 months
  0-15, higher means worse outcome

SECONDARY OUTCOMES:
uroflowmetry | 3 months
  curve shape
Frequency of void | 3 months
  defined as the number of voiding per day
International Prostate Symptom Score | 3 months
  0-35, with higher means worse outcome
EULAR Sjogren's Syndrome Patient Reported Index | 3 months
  0-30, with higher means worse outcome
Post-void residual | 3months
  the residual bladder volume after voiding, in mL
Average speed | 3months
  in ml/s, the average speed of voiding as measured by uroflowmetry

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan